CLINICAL TRIAL: NCT06791174
Title: Development and Validation of a Tumor Microenvironmental Collagen Signature Based on Multiphoton Imaging to Predict Superior Mediastinal Lymph Node Metastasis of Patients With Thyroid Cancer
Brief Title: Tumor Microenvironmental Collagen Signature to Predict Thyroid Cancer Superior Mediastinal Lymph Node Metastasis
Acronym: TC-CS-SMLNM
Status: Completed | Type: Observational
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Collaborators: Nanfang Hospital, Southern Medical University (Other); Sir Run Run Shaw Hospital (Other)
Responsible Party: Principal Investigator, Shumin Dong, Principal Investigator, The First Affiliated Hospital of Zhengzhou University
Other Study IDs: TC-TMECS-SMLNM-1.1
Record Dates: First submitted 2025-01-18; First posted 2025-01-24 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-01

CONDITIONS: Thyroid Cancer
Keywords: thyroid cancer; collagen; lymph nodes metastasis; predictive model; multiphoton imaging
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Paraffin tissue sections of primary tumor site
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- High TME Collagen Signature Group: The group with high tumor microenvironmental(TME) collagen signature. The TME collagen signature was developed in the training cohort and validated in external validation cohort and prospective cohort. The cutoff point of collagen signature was set according to the metastasis status of superior mediastinal lymph nodes.
- Low TME Collagen Signature Group: The group with low tumor microenvironmental(TME) collagen signature. The TME collagen signature was developed in the training cohort and validated in external validation cohort and prospective cohort. The cutoff point of collagen signature was set according to the metastasis status of superior mediastinal lymph nodes.

SUMMARY:
About 7-13% thyroid cancer patients have superior mediastinal lymph node metastasis, but its clinical identification is insufficient. Effective and individualized identification strategy need to be studied. Multiphoton imaging can accurately detect extracellular matrix collagen fibers by femtosecond laser. Quantitative features such as morphology and texture features extracted from the multiphoton images, can be used to predict lymph node metastasis of gastrointestinal cancer. Therefore, the investigators speculate that the characteristics of tumor microenvironment (TME) collagen based on multiphoton imaging may be used to predict superior mediastinal lymph node metastasis in thyroid cancer. The aim of this study is to investigate whether the TME collagen signature could predict superior mediastinal lymph nodes metastasis in thyroid cancer. The exposure of this observational cohort study is high TME collagen signature. The main measurement was the area under the receiver operating characteristic (AUROC) curves of collagen signature for predicting superior mediastinal lymph node metastasis.

DETAILED DESCRIPTION:
Retrospective cohorts were enrolled from the Sir Run Run Shaw Hospital of Zhejiang University School of Medicine, The First Affiliated Hospital of Zhengzhou University and Nanfang Hospital from January 2020 to December 2023. Perspective cohort was obtained from all the three centers from January 2024 to July 2024.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically diagnosed as thyroid cancer
* Radical surgery of tumor and simultaneous resection of superior mediastinal lymph nodes

Exclusion Criteria:

* Reoperation
* Under the age of 18
* Combined with thoracopathy, lymphoma or other diseases that may cause mediastinal lymph node enlargement
* The superior mediastinal lymph nodes metastasis status was not separately reported
* Insufficient pathology section quality
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with thyroid cancer
Sampling Method: Non-Probability Sample
Enrollment: 181 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Metastasis status of superior mediastinal lymph nodes | A week after operation generally
  Pathology result of superior mediastinal lymph nodes removed on the day of operation.

CONTACTS AND LOCATIONS:
Overall Officials: Shumin Dong (Princeple Investigator), M.D., Principal Investigator — The First Affiliated Hospital of Zhengzhou University; Detao Yin (Director of Thyroid Surgery Department), M.D., Study Director — The First Affiliated Hospital of Zhengzhou University
Locations (1):
- The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: Undecided